CLINICAL TRIAL: NCT00591942
Title: Outcome Evaluation of All Ceramic Crowns and Fixed Partial Dentures Bonded With Two Different Dental Cements.
Brief Title: Outcome Evaluation of Ceramic Crowns Using Two Different Dental Cements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clark Stanford (Other)
Responsible Party: Sponsor-Investigator, Clark Stanford, Associate Dean for Research & Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 200408065
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Sensitivity to Dental Cements; Dental Crowns; Dental Three-unit Bridges
Keywords: dental cement; ceramic crowns; three-unit bridges; sensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: 2 crowns per subject or one dental bridge with two retainer crowns for a total of 72 Teeth.
Who Masked: Participant
Masking Description: Subject unaware of the dental cement used on which crown or retainer
Oversight: Data Monitoring Committee: No

ARMS (2):
- VivaGlass dental cement (Active Comparator): 36 subjects (TOTAL) received two crowns each and another group of 11 subjects received a three-unit fixed dental bridge. Cross over design. One dental crown cemented with VivaGlass Cement/subject. Clinical visits to assess sensitivity and the integrity of the crowns/bridges occur at 6, 12, 18 and 24 months post seating of the restorations.
  Interventions: Device: Full ceramic crowns or 3-unit fixed partial dentures.
- MultiLink dental cement (Active Comparator): 36 subjects (TOTAL) received two crowns each and another group of 11 subjects received a three-unit fixed dental bridge. Cross Over design. One dental crown per subject was cemented with Multilink Dental Cement. Clinical visits to assess sensitivity and the integrity of the crowns/bridges occur at 6, 12, 18 and 24 months post seating of the restorations.
  Interventions: Device: Full ceramic crowns or 3-unit fixed partial dentures.

INTERVENTIONS:
Device: Full ceramic crowns or 3-unit fixed partial dentures. — Subjects who met the inclusion/excluson criteria received two ceramic crowns or one three-unit dental bridge on posterior teeth. The crowns and dental bridge were cemented using two different dental adhesives. Follow-up to assess sensitivity of the crowns/bridges occur at 24 hrs. and 1 week post seating by telephone. Clinical visits to assess sensitivity and the integrity of the crowns/bridges occur at 6, 12, 18 and 24 months post seating of the restorations.

SUMMARY:
The restoration of indirect partial and full coverage restorations in dentistry necessitates the use of a luting agent to act as a means of mechanical and potentially, chemical retention of the restoration. Upon the introduction of the first generation of glass Ionomer cements for use as a luting agent, an elevated short-term post operative hypersentivity was reported. In part, this adverse event was considered to be due to a desiccating effect of the cement as water is utilized in the setting reaction and thus a desiccation of the dentinal tubules was proposed as a potential mechanism leading to disruption of the neurosensory odontoblasts. Further materials development in the field of dental cement luting agents has lead to the introduction to the current market of resin formulations that have an alternative mechanism of setting. Consequently, there are anecdotal reports of a decrease in the incidence of post-operative sensitivity but no comparison with the effect of conventionally used dentin desensitizing agents as a part of the bonding process of the restoration.

The purpose of this trial is a single blinded parallel design randomized clinical trial to evaluate the perceived incidence of post-operative sensitivity when full coverage all ceramic crowns or short-span three unit fixed partial dentures (dental bridge) is fabricated in the posterior part of the mouth. The dental crowns or bridges will be bonded with conventional glass ionomer cement or a Urethane dimethacrylate / Bis-GMA composite resin dental cement. Outcome measures will be both objective clinical criteria and the use of a calibrated pain survey instrument.

DETAILED DESCRIPTION:
Background and Significance: The development of porcelain crowns for the predictable restoration of teeth has been brought about by the development of bonding techniques to enamel and dentin with the use of multi-step total etch adhesive systems along with the evolution in small particle hybrid resin composites as adhesive luting agents. One of the most common post-operative concerns of patients following delivery of full coverage crowns and bridges is sensitivity to thermal conditions in the mouth (cold water, ice cream, etc.) (Goodacre, Bernal et al. 2003). In order to understand the biological basis for these materials it is important to understand the anatomy and neurophysiology of dentin. The following is adapted from a paper provided by Dr. Charles Cox (Professor, University of Alabama School of Dentistry) concerning dentin structure and mechanisms for reduction of dentin hypersensitivity .

Dentin is a vital tissue, harder than bone but weaker than enamel with a physiological elasticity preventing tooth fracture. Dentin is approx. 74% mineral; the organic phase being approx. 26% type-1 collagen with small amounts of proteins and water. The collagen matrix is secreted as a biologically "plastic" material, which hardens by a variety of mechanisms. Normal dentin is composed of millions of tubules or canals, running from the pulpal wall to the Dentin-Enamel Junction (DEJ). The dimensions of these tubules or canals varies depending on the position within the dentin structure. For instance, tubule diameter at the DEJ is 0.06 µm, and 3.0 µm at the pulpal wall (approx. 60,000 tubules / mm2). Most tubules are filled with fluid, an odontoblast cell process, collagen, and occasional non-myelinated pulpal nerves coursing approx. 150 µm towards the DEJ (Ten Cate 1998).

In normal (non-anesthetized) patients, Gysi (1900) reported that fluid distortion on the cavity floor caused sharp pain. Brännström et al. (1966, 1969, 1976, 1979, 1980, 1996) demonstrated dentin hypersensitivity (sharp pain) is the result of rapid fluid movement in the tubule complex, aggravated by aggressive air-drying. Physiological testing in various animal studies (Heyeraas 1985, Narhi 1983, 1985) confirmed the fluid pulsing or hydrodynamic mechanism (Brännström 1966) as the prime cause of sudden dentin pain. Physiologically, any rapid bi-directional fluid flow is the result of a sudden shift in tubule fluid from stimuli (i.e. cold or rapid airflow; Brännström 1996).

Management of dentin hypersensitivity is only one part of a successful dental complete coverage restoration (dental crown or bridge). In evaluating the clinical service-life of porcelain crowns there are three aspects of the bonding environment that needs to be considered. These consist of the tooth preparation, the adhesive and the tooth or crown preparation and the fit of the porcelain restoration to the tooth preparation. All ceramic restorations need enamel and dentin reduction of at least 1.5 mm along with a smooth shoulder and avoidance of sharp edges to avoid crack formation on the intaglio surface, proper esthetics, physiological contours and strength of the final restoration.(Goodacre, Campagni et al. 2001) Dental preparation for full coverage restorations (1.5 to 2 mm clearance which often means 1.5 - 2 mm loss of tooth structure) are inherently non-conservative and with a reduced amount of remaining tooth structure there is an elevated risk of post-operative sensitivity.

In today's society, having a dental restoration that provides minimal post-operative sensitivity is only part of the demand from patients. There is an increasing expectation for esthetic, "life-like" restorations that simulate if not replicate the natural tooth. This is complicated especially in patients with heavy occlusion or are missing teeth. The development of CAD/CAM milling technologies has laid the groundwork for use of high strength heat-pressed zirconia [tetragonal zirconia polycrystals (TZP) a yttrium partially stabilized polycrystal structure] as a supporting framework for supporting an esthetic, "life-like" Lucite-base veneering ceramic material to provide an all ceramic form of full coverage dental restorations for individual teeth or replacement of a single missing tooth with a 3-united fixed partial denture ("dental bridge"). The use of press porcelain crown technology has allowed the improvement of fit of refractory die porcelain crown fabrication relative to conventional Pt foil techniques and may lead to greater predictability and reduced microleakage (with enhanced service life of the dental restoration). The potential for an enhanced service life may depend on a combination of silination with a bifunctional bis-GMA primer and dual cured composite resin luting agent which may seal microcracks within the intaglio surface of the porcelain and a sufficient bond to tooth structure for a reasonable service life.

ELIGIBILITY:
Inclusion and Exclusion Criteria:

* Subject shall be in need of a maximum of two porcelain crowns on their posterior teeth. In the case of missing single teeth, the adjacent retainers shall be in need of complete coverage restorations and provide sufficient support for a conventional 3-unit fixed partial denture.
* Cantilever pontics shall not be performed.
* Prospective teeth shall be vital and not in need of root canal endodontic therapy.
* The tooth in question shall be "responsive" to conventional Endodontic tests. These tests shall include a positive response to thermal stimulation (CO2 ice) and/or electric pulp testing (EPT).
* The tooth in question shall be in occlusion with the opposing dentition. Subjects shall have an Angle Class I occlusion with preferably canine eccentric lateral guidance. In selected cases a mutual protected occlusion is acceptable if lateral guidance can be minimized on the restorations at risk. Subjects with intraoral ornamental metallic devices (e.g., posts, etc) shall be excluded.
* The tooth in question shall not be a retainer for a Removable Partial Denture (i.e., a surveyed crown) although the tooth may lack a mesial or distal contact.
* The tooth in question shall have periodontal stability (probing depths < 3mm, dental mobility < 1).
* The tooth shall not be in need of surgical crown lengthening for reasons of restoration or periodontal status.
* Subjects involved in other clinical trial protocols utilizing a similar protocol as proposed shall be excluded.
* The subject shall not have any known allergies to any materials used in this protocol. Subjects who need antibiotic prophylaxis for SBE are acceptable for inclusion.
* Subjects of child bearing age shall have a urine pregnancy test. Pregnant subjects shall be excluded.
* Subjects shall be available for a potential recall period of five years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clark Stanford, DDS, PhD, Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa College of Dentistry, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
IPD data is tied to Hippa identifiers and therefore cannot be released

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects needing a dental crown or dental bridge
Units Other Than Participants: Crowns
Groups:
- VivaGlass Cement: Cross over design, two crowns per subject, one crown cemented with VivaGlass/subject
- Multilink Cement: Cross over design, two crowns per subject, one crown cemented with Multilink/subject
Period: Overall Study
Arm/Group | VivaGlass Cement | Multilink Cement
Started (Participants enrolled in both arms. 2 teeth were used in each subject, each with differing cement.) | 36; 36 Crowns | 36; 36 Crowns
Completed | 36; 36 Crowns | 36; 36 Crowns
Not Completed | 0; 0 Crowns | 0; 0 Crowns

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Note only one group is listed since EACH subject received TWO crowns. AS cross-over design, ONE crown had the VivaGlass cement and the second crown (in the same subject) had the Multi-link cement.
Arm/Group | Group 1
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Post-operative Pain (Yes/no)
Description: Scores reported are subjects reporting any pain (yes/no)
Time Frame: Outcome is measured: 24 hrs., 7 days, and 6, 12, 18 and 24 months following seating of the restorations
Measure: Number; unit: participants
Units Other Than Participants: crowns
Groups:
- Ivoclar Vivaglass CEM IC Cement: Ivoclar Vivaglass CEM IC cement for ceramic crowns and 3-unit dental bridge
- Ivoclar/Vivadent Composite Resin Cement: Ivoclar/Vivadent Composite Resin Cement for ceramic crowns and 3-unit dental bridge
Arm/Group | Ivoclar Vivaglass CEM IC Cement | Ivoclar/Vivadent Composite Resin Cement
Number analyzed (Participants) | 36 | 36
Number analyzed (crowns) | 36 | 36
participants
  0 Hour | 1 | 0
  24 hours | 1 | 2
  7 days | 3 | 5
  6 month | 4 | 3
  12 months | 2 | 3
  18 months | 3 | 3
  24 months | 3 | 3
Statistical Analysis 1: Comparison: Ivoclar Vivaglass CEM IC Cement vs Ivoclar/Vivadent Composite Resin Cement; Test type: Non-Inferiority — 95% CI were used; p = 0.5637, Chi-squared; df=1; KM Survival Curves = 0.5637

ADVERSE EVENTS:
Time Frame: 0 to 24 months
Description: side effects of the dental procedures from transient pain to intervention. All patient and clinician reported side effects was recorded.
Groups:
- Ivoclar Vivaglass CEM IC: Ivoclar Vivaglass CEM IC cement for ceramic crowns and 3-unit dental bridge
- Ivoclar/Vivadent Composite Resin: Ivoclar/Vivadent Composite Resin Cement for ceramic crowns and 3-unit dental bridge
Arm/Group | Ivoclar Vivaglass CEM IC | Ivoclar/Vivadent Composite Resin
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 1/36 | 0/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivoclar Vivaglass CEM IC (N=36) | Ivoclar/Vivadent Composite Resin (N=36)
Crown Fracture (General disorders) | 1 (1) | 0 (0) — Crown Fracture

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No